CLINICAL TRIAL: NCT06728098
Title: Safety and Tolerability Evaluation of Heat-Inactivated Akkermansia Muciniphila Akk11: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Safety and Tolerability Evaluation of Akkermansia Muciniphila
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WK2024017
Record Dates: First submitted 2024-11-27; First posted 2024-12-11 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2024-10

CONDITIONS: Healthy
MeSH Terms: interventions — Probiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Live Akk11 (Experimental): Healthy Subjects Receiving Probiotic live Akk11: One probiotic Akkermansia muciniphila Akk11 capsule daily (30 billion AFU/capsule).
  Store in cool and dry place, without exposure to light.
  Interventions: Dietary Supplement: Probiotic
- Inactivated Akk11 (Experimental): Healthy Subjects Receiving Probiotic Inactivated Akk11: One probiotic Akkermansia muciniphila Akk11 capsule daily (30 billion TFU/capsule).
  Store in cool and dry place, without exposure to light.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Healthy Subjects Receiving Placebo : Take 1 maltodextrin capsule every day. Store in cool and dry place, without exposure to light.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Probiotic — The experimental phase of this study had last 30 days and each patient will make 3 visits (d1,d15,d30).
  Arms: Inactivated Akk11; Live Akk11
Dietary Supplement: Maltodextrin — The experimental phase of this study had last 30 days and each patient will make 3 visits (d1,d15,d30).
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded, placebo-controlled study to evaluate the efficacy and safety of Akkermansia muciniphila Akk11 in healthy adult.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subject age 18-60 years at screening.
2. Healthy subject according to investigator judgement based on screening data.
3. Subjects must be either of non-childbearing potential, or if of childbearing potential, they must be abstinent or have practiced adequate contraception for the entire study.
4. Subjects who have not smoked in the past 1 month prior to screening.
5. Subjects with a healthy and balanced diet, including adequate fiber intake in their food consumption.
6. Subject or subject's legally acceptable representatives have the ability to comply with the trial protocol.
7. Signed informed consent from the subject or subject's legally acceptable representatives (must be obtained before any trial related activities).

Exclusion Criteria:

1. History of or presence of diabetes, immunodeficiency disorders, or chronic illness.
2. Regular use of medications known to affect the gastrointestinal system or alter gut microbiota composition, including but not limited to antibiotics, and immunosuppressants.
3. Have continuous, daily use of probiotics or probiotic containing products within 1 month prior to randomization.
4. Pregnant, planning a pregnancy or lactating female (urinary pregnancy test will be applied to female subjects at screening).
5. Change type of diet during study.
6. Any known allergy or intolerance to any of the ingredients in the formulation of the product under study.
7. History of drug, alcohol or other substance abuse, or other factors that limit their ability to cooperate during the study.
8. History of or presence of eating disorder.
9. Subject whose condition does not make them eligible to the study, according to the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Changes in stool quality | 30 days
  Stool consistency (using the Bristol Stool Scale) from baseline to day 30. The Bristol Stool Scale is a tool to assess gut health by classifying feces into seven categories based on shape and consistency: types 1-2 indicate constipation, 3-4 are normal, and 5-7 suggest diarrhea.

CONTACTS AND LOCATIONS:
Locations (1):
- Fakultas Kedokteran Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia